CLINICAL TRIAL: NCT00215904
Title: D-serine Adjuvant Treatment for Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Princepal Investigator, Herzog Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: Heresco1CTIL; 20030312
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: D-serine (~2g/day)
- 2 (Experimental)
  Interventions: Drug: D-serine (~2g/day)

INTERVENTIONS:
Drug: D-serine (~2g/day) — Two 6 weeks treatment arms. One arm: adjuvant treatment with D-serine (~2g/day). Second arm : adjuvant treatment with placebo (~2g/day).

SUMMARY:
The proposed experiment will evaluate the effects of the NMDA receptor full agonist D-serine (~2g/day) on persistent symptoms of Parkinson's Disease and on antiparkinsonian drugs-induced dyskinesias.

D-serine will be used as add-on therapy to on-going medications received by Parkinson's Disease patients. The rational for this study stems from observations made in pervious clinical trials with schizophrenia patients, in which it was demonstrated that D-serine adjuvant treatment resulted in:1)improvement of parkinsonian side effects induced by antipsychotic drugs and 2) improvement of depression and negative (i.e apathy, blunted effects, anhedonia) symptoms which are similar to symptoms encountered in Parkinson's Disease.

The study will have a crossover design in accordance to which each patient will receive, in random order D-serine and placebo for a 6 weeks period each. Thus, any participant will have the opportunity to receive the experimental treatment.

ELIGIBILITY:
Inclusion Criteria:

* PD diagnosis
* ≥2 on UPDRS items 32,33
* receive treatment with L-dopa alone or in combination with other antiparkinsonian medications.

Exclusion Criteria:

* current or previous history of other neurological disorders
* unstable medical conditions
* renal pathology
* pregnant female patients excluded

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
UPDRS scores | 6 weeks
PANSS scores | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, Principal Investigator — Ezrath Nashim - Herzog Memorial Hospital
Locations (1):
- Ezrath Nashim - Herzog Memorial Hospital, Jerusalem, Israel

REFERENCES:
- [Derived] Gelfin E, Kaufman Y, Korn-Lubetzki I, Bloch B, Kremer I, Javitt DC, Heresco-Levy U. D-serine adjuvant treatment alleviates behavioural and motor symptoms in Parkinson's disease. Int J Neuropsychopharmacol. 2012 May;15(4):543-9. doi: 10.1017/S1461145711001015. Epub 2011 Jul 7. PMID 21733283